CLINICAL TRIAL: NCT04151199
Title: Molecular Transducers of Physical Activity Consortium (MoTrPAC) - Pediatric Protocol
Acronym: MoTrPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Stanford University (Other); Broad Institute of MIT and Harvard (Other); Duke University (Other); Emory University (Other); Icahn School of Medicine at Mount Sinai (Other); Mayo Clinic (Other); Pacific Northwest National Laboratory (U.S. Federal Agency); University of Michigan (Other); Wake Forest University (Other); University of Vermont (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00057366; U01AR071158 (NIH); U24AR071113 (NIH); U24OD026629 (NIH); U24DK112349 (NIH); U24DK112342 (NIH); U24DK112340 (NIH); U24DK112341 (NIH); U24DK112326 (NIH); U24DK112331 (NIH); U24DK112348 (NIH)
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-05

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The randomized trial is conducted in accordance with an intent-to-treat (ITT) design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Intervention Control (No Intervention): The control group is randomized but does not participate in the intervention but does complete the acute test and biospecimen collection following the intervention period.
- Endurance Exercise (Active Comparator): Participants randomized to EE participate in the intervention and complete the acute test and biospecimen collection following the intervention period.
  Interventions: Other: EE Training
- Cross Sectional HA (No Intervention): Do not participate in intervention after single acute exercise test of Endurance Exercise.
- Cross Sectional LA (No Intervention): Do not participate in intervention after single acute exercise test of Endurance Exercise.

INTERVENTIONS:
Other: EE Training — Participants randomized to EE training engage in three school-based or center-based (PERC) EE training sessions each week for approximately 12 weeks; each session lasting roughly 70 min with a 45-50 minutes of a stimulus phase and the remaining time being used to warm-up and cool down.
  Arms: Endurance Exercise

SUMMARY:
The goal of the Molecular Transducers of Physical Activity Consortium (MoTrPAC) is to assess molecular changes that occur in response to physical activity (PA). To achieve this aim, studies will be conducted in adults and separately in children and adolescents. The UC Irvine MoTrPAC Pediatric Clinical Center oversees two interrelated study phases in children and adolescents:

1. A cross-sectional phase in which molecular transducers (obtained from blood sampling) are measured in response to an acute exercise challenge (n = 320);
2. An intervention phase is conducted as a mechanistic randomized controlled trial (RCT). Participants are recruited from the cross-sectional study phase and randomized to endurance exercise (EE) training (n = 120) or no exercise Control (n = 50) for a period of approximately 12 weeks.

DETAILED DESCRIPTION:
The overarching hypothesis is that there are discoverable molecular transducers that communicate and coordinate the effects of exercise on cells, tissues, and organs, which may initiate processes ultimately leading to the health benefits of exercise. Because this is a mechanistic trial, the main goal is not a single health-related outcome. Rather, the goal is to generate a resource leading to the generation of a map of the molecular responses to exercise that will be used by the Consortium and by the scientific community at large to generate hypotheses for future investigations of the health benefits of PA. Study assessments are completed before and after the intervention period (exercise or control), and at specific interim time points during the intervention. An additional focus of the pediatric studies is to examine the impact of sex and developmental phase (self-reported pubertal stage) during childhood and adolescence on acute and chronic exercise responses.

Assessments include measurements of cardiorespiratory fitness, muscular strength, and body composition (including whole body bone mineral content) determined by dual-energy x-ray absorptiometry (DXA). There is also collection of blood, monitoring of free-living PA level using wearable devices, and completion of participant reported outcomes and health status by interview and/or questionnaire. As part of the MoTrPAC functions, participant data and biological samples are transferred from the Pediatric Clinical Site to the Consortium Coordinating Center (CCC) Data Management, Analysis and Quality Control Center (DMAQC) and to the Biological Sample Repository, and later analyzed by the Consortium Chemical Analysis Sites (CAS) and the Bioinformatics Center (BIC).

Biological samples collected in this project undergo molecular phenotyping, including metabolomic, lipidomic, proteomic, epigenomic, transcriptomic, and genomic analyses. These assays are done at the MoTrPAC CAS.

Overall coordination of the study and analyses occurs at 4 institutions which make up the CCC and the BIC.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian and participant are willing to provide informed consent and assent to participate in the MoTrPAC Study
* Must be able to read and speak English well enough to provide informed consent, assent and understand instructions
* Children and adolescents ages 10-17 (Pubertal stages 1-5)
* Determined to be in good health by pre-participation medical history review performed at PERC
* BMI %ile (>5th, <95th)
* Weight ≥30 Kg (minimum required for blood collection)
* LAEE children defined as self-reported of no more than 2 days per week, lasting no more than 120 minutes per week, of regular (structured) intense endurance exercise (e.g., running, cycling, elliptical, soccer, swimming and rowing activity that results in feelings of substantially increased heart rate and rapid breathing and sweating with limited ability to talk) in the 3 months prior to study enrollment.
* HAEE children in this study is defined as:
* self-reported participation in a structured/regular endurance sports (e.g., running, cycling, soccer, swimming and rowing activity that results in feelings of substantially increased heart rate and rapid breathing and sweating with limited ability to talk).
* Participation in these activities is ≥4 times per week (>240 min per week) for at least 9 months prior to study enrollment.

Exclusion Criteria:

* Self-report or laboratory evidence of familial hyperlipidemia/dyslipidemia (e.g., total cholesterol ≥ 200mg/dL and or triglyceride ≥ 100mg/dL)
* Daily or weekly chronic use of any prescription medication in the past 3 months (excluding birth control)
* Any use of tobacco, e-cigarettes, illegal drugs, alcohol, or marijuana (self-report) within the last 12 months
* Pregnancy or breastfeeding
* Sudden or abrupt (≥5%) weight lost (self-report) over the preceding 3 months
* Past history of serious chronic diseases (including, but not limited to: asthma, diabetes, juvenile idiopathic arthritis, cystic fibrosis, malignancy, congenital heart disease, cerebral palsy, muscular dystrophy, autoimmune diseases, inflammatory bowel disease)
* Evidence of disease, disability or other condition that would impair participation in physical activity as determined by a study clinician
* Blood donation in the past 3 months (self-report)

Similar inclusion/exclusion criteria are being used for the intervention phase, with the additional exclusion criterion of children who meet the definition of HAEE defined above.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
CPET VO2 Peak | Baseline; Week 12
  Changes in CPET VO2 Peak calculated as L/min
Isometric Knee Peak Torque by Group | Baseline; Week 12
  Changes in peak torque measured in Newton Meters

SECONDARY OUTCOMES:
HDL-C | Baseline; Week 12
  Changes in HDL-C (mg/dL)
LDL-C | Baseline; Week 12
  Changes in LDL-C (mg/dL)
Triglycerides | Baseline; Week 12
  Changes in Triglycerides (mg/dL)
HbA1C | Baseline; Week 12
  Changes in HDL-C (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Mike E Miller, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared publically through the MoTrPAC data hub based on the consent and assent choices of the parent/participant. PHI will not be released.
Supporting Information: Study Protocol
Time Frame: The timeframe for data sharing is unknown at this time. Estimated time for release is end of 2026.
Access Criteria: All data and supporting information will be made available through the MoTrPAC Data Hub (https://motrpac-data.org/). Data Access can be requested and public repositories will be outlined on the data hub website.
URL: https://motrpac-data.org/

REFERENCES:
- [Background] MoTrPAC Study Group; Jakicic JM, Kohrt WM, Houmard JA, Miller ME, Radom-Aizik S, Rasmussen BB, Ravussin E, Serra M, Stowe CL, Trappe S, Abouassi H, Adkins JN, Alekel DL, Ashley E, Bamman MM, Bergman BC, Bessesen DH, Broskey NT, Buford TW, Burant CF, Chen H, Christle JW, Clish CB, Coen PM, Collier D, Collins KA, Cooper DM, Cortes T, Cutter GR, Dubis G, Fernandez FM, Firnhaber J, Forman DE, Gaul DA, Gay N, Gerszten RE, Goodpaster BH, Gritsenko MA, Haddad F, Huffman KM, Ilkayeva O, Jankowski CM, Jin C, Johannsen NM, Johnson J, Kelly L, Kershaw E, Kraus WE, Laughlin M, Lester B, Lindholm ME, Lowe A, Lu CJ, McGowan J, Melanson EL, Montgomery S, Moore SG, Moreau KL, Muehlbauer M, Musi N, Nair VD, Newgard CB, Newman AB, Nicklas B, Nindl BC, Ormond K, Piehowski PD, Qian WJ, Rankinen T, Rejeski WJ, Robbins J, Rogers RJ, Rooney JL, Rushing S, Sanford JA, Schauer IE, Schwartz RS, Sealfon SC, Slentz C, Sloan R, Smith KS, Snyder M, Spahn J, Sparks LM, Stefanovic-Racic M, Tanner CJ, Thalacker-Mercer A, Tracy R, Trappe TA, Volpi E, Walsh MJ, Wheeler MT, Willis L. Molecular Transducers of Physical Activity Consortium (MoTrPAC): human studies design and protocol. J Appl Physiol (1985). 2024 Sep 1;137(3):473-493. doi: 10.1152/japplphysiol.00102.2024. Epub 2024 Apr 18. PMID 38634503

DOCUMENTS (1):
  • Informed Consent Form (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT04151199/ICF_000.pdf